CLINICAL TRIAL: NCT04898660
Title: The Role of the Embedded Participant on Learners' Performance During High- Fidelity Simulation
Brief Title: The Embedded Participant During High-fidelity Simulation
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Other Study IDs: FAC1
Record Dates: First submitted 2021-05-10; First posted 2021-05-24 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: High Fidelity Simulation; Simulation Training/methods; Task Performance and Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Simulation in medicine is a powerful and effective teaching tool that has become essential for the training of students and health professionals.

In this context, simulation instructor training have been implemented in recent years, where many subjects are addressed, such as the main principles of pedagogy, the integration of simulation, the construction of a scenario, briefing and debriefing.

However, scenario facilitation, in particular the role of the embedded participant (EP), is only vaguely discussed. The EP of a high-fidelity simulation session plays a very important role in driving the scenario. Indeed, he/she guides the learner in order to achieve all the educational objectives set by the main instructor of the scenario. He/she also manages unexpected behavior and possible technical issues that may arise. Finally, the EP supervises the physical and psychological risks inherent in the simulation in order to maintain a safe environment.

All of these key roles suggest that the EP can influence the performance of the learners. Little is known about the relationship between Facilitation and Learner Performance.

In this observational study, investigators aim to explore the influence of the embedded participant on learners' technical and non-technical performances during high-fidelity simulation by analysing previously recorded sessions.

DETAILED DESCRIPTION:
In this observational study, investigators aim to measure performance on high-fidelity simulation scenarios (HFS) used routinely in the current anesthesiology, training curriculum. Age, sex, previous experience of HFS will be noted. All data will be anonymized.

Two investigators will independently evaluate the performance of HFS by video record:

* technical performance on tables pre-established by experienced instructors and based on international recommendations,
* non-technical performances, assessed using the Ottawa Global Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Resident physicians in anesthesia/intensive care- postgraduate year 1-5 participating in HFS training sessions from 2015 to 2021
* Consent for recording

Exclusion Criteria:

* Denial to be recorded

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anaesthesia residents in postgraduate years 1-5 at Edouard Herriot Hospital, Lyon
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Technical Skills Performance | 1 month (review video)
  technical performance on a scale pre-established according to each scenario rated from 0 to 100.
Non-technical skills performance | 1 month (review video)
  Ottawa Crisis Resource Management Global Rating Scale rated from 6 to 42.

SECONDARY OUTCOMES:
Demographic characteristics | 1 month (collect data)
  demographic data related to the instructors (embedded participants) through a questionary

CONTACTS AND LOCATIONS:
Overall Officials: thomas rimmele, PhD, Study Chair — Claude Bernard University
Locations (1):
- Claude Bernard University, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooke JM, Rooney DM, Fernandez GL, Farley DR. Simulation center best practices: A review of ACS-accredited educational institutes' best practices, 2011 to present. Surgery. 2018 Apr;163(4):916-920. doi: 10.1016/j.surg.2017.11.004. Epub 2017 Dec 19. PMID 29273177
- [Background] Paige JB, Graham L, Sittner B. Formal Training Efforts to Develop Simulation Educators: An Integrative Review. Simul Healthc. 2020 Aug;15(4):271-281. doi: 10.1097/SIH.0000000000000424. PMID 32218086
- [Background] Lewis KL, Bohnert CA, Gammon WL, Holzer H, Lyman L, Smith C, Thompson TM, Wallace A, Gliva-McConvey G. The Association of Standardized Patient Educators (ASPE) Standards of Best Practice (SOBP). Adv Simul (Lond). 2017 Jun 27;2:10. doi: 10.1186/s41077-017-0043-4. eCollection 2017. PMID 29450011
- [Background] Boyer TJ, Mitchell SA. Utilization of Embedded Simulation Personnel in Medical Simulation. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK562294/ PMID 32965965